CLINICAL TRIAL: NCT04474171
Title: An Online Self-management Program for Spinal Cord Injury: Feasibility Study of SCI&U
Acronym: SCI&U
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Susan Jaglal, Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 505419; 399095 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCI&U Intervention (Experimental): The SCI&U online platform has a resource library, secure videoconferencing, and tools to support one-on-one health coaching. Health coaches are certified in motivational interviewing and have lived in the community with SCI for more than five years. In the first session, participants identify priority issues related to their health and target management of secondary conditions specific to SCI. They will work through goal setting, problem solving activities and create action plans for behaviour change, which will be securely stored. The intervention will be a maximum of 14 sessions over 6 months. Each session will cover a health-related topic (bladder, bowel, skin, pain, healthy eating, physical activity or stress, anxiety and depression) and a self-management skill topic (action planning, goal setting, problem-solving, mood management, navigating the health care system and communicating with health care providers) with an expected duration of 30 to 45 minutes.
  Interventions: Behavioral: SCI&U online health coaching program
- Waitlist Control (No Intervention): Usual health care and be offered the SCI&U program at the end of the 12-month follow-up period (wait-list control)

INTERVENTIONS:
Behavioral: SCI&U online health coaching program — Online secure videoconferencing health coaching platform with resource library to promote self-management. Maximum number of sessions is 14 over 6 months and covers health related topics to reduce secondary complications
  Arms: SCI&U Intervention

SUMMARY:
Managing a spinal cord injury (SCI) is a life-long process. Within the first year of injury, more than 50% of people discharged with a SCI may require re-hospitalization due to a secondary complication, such as a urinary tract infection, pressure ulcer or pneumonia. Even 20 years post-injury, re-hospitalization rates remain over 30%. While re-hospitalization rates in Canada have remained high for more than 10 years, the length of stay in inpatient rehabilitation has decreased dramatically, thereby limiting the time for provision of health information and skill acquisition in the inpatient rehabilitation setting. There is growing evidence from two recent pilot trials to suggest that self-management programs that provide appropriate health information, skills and telephone-based support for community-dwelling patients with SCI improves health behaviors and leads to reductions in re-hospitalization.

Goals/Research Aim: To conduct a pilot RCT (feasibility study) that will inform the design of a definitive RCT to determine whether an online self-management program incorporating trained peer health coaches (called "SCI&U") compared to usual care will result in improved self-management skills (short-term outcome) and lead to reduced days of hospitalization (long-term outcome) due to secondary complications.This pilot study is a two-group RCT with an embedded qualitative component. The target population is adults with SCI who have been discharged from inpatient rehabilitation and living in the community. Sixty subjects will be recruited from across Canada with a focus on British Columbia and Ontario and randomly assigned to the SCI&U intervention or usual care.

Evaluations will occur at baseline, 2, 6, and 12 months.

DETAILED DESCRIPTION:
Background and Importance: Managing a spinal cord injury (SCI) is a life-long process. Within the first year of injury, more than 50% of people discharged with a SCI may require re-hospitalization due to a secondary complication, such as a urinary tract infection, pressure ulcer or pneumonia. Even 20 years post-injury, re-hospitalization rates remain over 30%. While re-hospitalization rates in Canada have remained high for more than 10 years, the length of stay in inpatient rehabilitation has decreased dramatically, thereby limiting the time for provision of health information and skill acquisition in the inpatient rehabilitation setting. There is growing evidence from two recent pilot trials to suggest that self-management programs that provide appropriate health information, skills and telephone-based support for community-dwelling patients with SCI improves health behaviors and leads to reductions in re-hospitalization.

Goals/Research Aim: To conduct a pilot RCT (feasibility study) that will inform the design of a definitive RCT to determine whether an online self-management program incorporating trained peer health coaches (called "SCI&U") compared to usual care will result in improved self-management skills (short-term outcome) and lead to reduced days of hospitalization (long-term outcome) due to secondary complications.

Secondary outcomes include self-efficacy for self-management, depression, resilience, number and severity of secondary conditions, health-related quality of life, and patient-reported unplanned ED visits.

Methods/Approaches/Expertise: This pilot study is a two-group RCT with an embedded qualitative component. The target population is adults with SCI who have been discharged from inpatient rehabilitation and living in the community. Sixty subjects will be recruited from across Canada with a focus on British Columbia and Ontario and randomly assigned to the SCI&U intervention or usual care.

Evaluations will occur at 0, 2, 6, and 12 months. At 6 and 12 months, interviews will be conducted with SCI&U participants and at 12 months focus groups with health coaches, consumer organizations, and rehabilitation hospital staff to explore the feasibility of the study protocol, understand perceived costs and benefits of SCI&U, and sustainability considerations. The creation of the SCI&U online self-management program is based on a number of studies conducted by the research team. The investigators initially determined implementation considerations in terms of need, content and mode of delivery in a mixed methods study of individuals with SCI, their family members, and hospital managers. The SCI&U team includes rehabilitation researchers, persons with SCI, community-based organizations (SCI BC, SCI Ontario and Praxis Spinal Cord Institute) and clinicians from across Canada. The investigators used an integrated knowledge translation approach where users with SCI co-designed and developed the prototype. The investigators have completed usability testing on 20 participants and trained 5 health coaches and had an additional 11 individuals living with SCI complete 6 sessions of health coaching using the SCI&U prototype.

Expected Outcomes: The findings from this feasibility study are integral to the development of a definitive RCT. It is anticipated that SCI&U would not only reduce secondary complications and subsequent inappropriate health care use, but also improve the quality of life for individuals with SCI.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 6 months post-injury to allow time to adjust to injury;
2. living in the community;
3. age ≥18 years;
4. ability to speak and read English and
5. have a primary care physician

Exclusion Criteria:

1. currently participating in another formal self-management program and
2. self-report of physician diagnosed concurrent traumatic brain injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Skill and Technique Acquisition Scale from the Health Education Impact Questionnaire | 6 and 12 months after baseline
  4-item scale that captures knowledge based skills and techniques that persons acquire to help them cope with health problems. It is a 4-point Likert scale (1-4) ranging from strongly disagree to strongly agree. Score is the sum of the 4 items. A higher score means a better outcome.
Health Care Utilization: Cumulative days re-hospitalized 12 months after baseline | 12 months after baseline
  Self-report of total days hospitalized for each participant will be obtained as the primary health care utilization outcome. This will be measured at 6 and 12 months after baseline with the qeustion "how many total NIGHTS did you spend in the hospital in the past 6 months? A higher total number of days means a worse outcome.

SECONDARY OUTCOMES:
Secondary Conditions Scale | 6 and 12 months after baseline
  This is a 16-item self report measure that targets secondary conditions associated with SCI that impact health. The response options are a 4-point scale (0 - not experienced in the last 3 months or is an insignificant problem, 1 mild or infrequent problem, 2 moderate or occasional problem, 3 significant or chronic problem. Score is the sum of the 16 items. A higher total score means a worse outcome.
University of Washington Self-Efficacy Scale for People with Disabilities and Chronic Conditions: Short Form | 6 and 12 months after baseline
  6-item self-report questionnaire rating confidence in self-management skills on a 5-point Likert scale ranging from "0" not at all to '4" completely. Score is the sum of the 6 items. A higher score means a better outcome (self-efficacy).
International Spinal Cord Injury Datasets Quality of Life Basic Dataset-Data Form (Version 1.0) | 6 and 12 months after baseline
  3 questions from the International SCI QOL Basic dataset that rates satisfaction with general QOL, physical and psychological health on an 11-point Likert scale with "0" being completely dissatisfied" to '10" completely satisfied. A higher score means a better outcome.
SCI-QOL Resilience Short Form | 6 and 12 months after baseline
  8-item measure of adaptation or adjustment after the injury. The context for all resilience items is "in the past 7 day...". The response options are a 5-point Likert scale ranging from "1" Never to "5" Always. Score is the sum of the 8 items. A higher score means a better outcome.
Personal Health Questionnaire Depression Scale (PHQ-8) | 6 and 12 months after baseline
  8-item Likert scale measuring depression symptoms. Response options range from "0" not at all to "3" nearly every day. Score is the sum of the 8 items. A higher score means a worse outcome. A score of 10 or greater is considered major depression, 20 or more is severe major depression symptoms.
Self-reported Emergency department visits | 6 and 12 months
  self-report number of emergency department visits in the past 6 months. The question is "In the past 6 months, how many times did you go to a hospital emergency room?" A higher number indicates more visits and means a worse outcome
Social/Role Activities Limitations | 6 and 12 months after baseline
  4-item self-report measure of limitations within the past 2 weeks. This is scored on a 5-point Likert scale with "0" as not at all and '4" almost daily. The score of the scale is he mean of the four items. A higher scores indicates greater activities limitations.
Positive and Active Engagement in Life from the Health Education Impact Questionnaire | 6 and 12 months after baseline
  5-item scale assesses motivation to be active and engaging in life-fulfilling activities as a result of self-management program involvement
Self Monitoring and Insight from the Health Education Impact Questionnaire | 6 and 12 months after baseline
  6-item scale captures the individuals' ability to monitor their condition, and their physical/emotional responses that lead to insights and actions to self manage
Health Services Navigation from the Health Education Impact Questionnaire | 6 and 12 months after baseline
  5-item scale captures individual's understanding of and ability to interact with health professionals and confidence and ability to communicate and negotiate to get needs met
Emotional Distress from the Health Education Impact Questionnaire | 6 and 12 months after baseline
  6-item scale measures overall negative affective responses to illness including anxiety, anger, and depression

CONTACTS AND LOCATIONS:
Overall Officials: Susan B Jaglal, PhD, Principal Investigator — Professor
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
aggregated data from descriptive and outcomes measures will be shared
Supporting Information: Study Protocol, ICF
Time Frame: after publication of main study manuscript and for 5 years
Access Criteria: need permission from PI

REFERENCES:
- [Derived] Jaglal SB, Allin SJ, Craven BC, Guilcher SJT, Linassi AG, McBride CB, Moineddin R, Mortenson WB, Munce S, Salbach NM, Shepherd JD, Sweet SN, Thorson T, Tomasone JR. A pilot randomised controlled trial of the Spinal Cord Injury and You (SCI&U) online peer health coaching self-management program. Pilot Feasibility Stud. 2026 Jan 28. doi: 10.1186/s40814-026-01769-y. Online ahead of print. PMID 41593819